CLINICAL TRIAL: NCT01155752
Title: Z4770s, Use of Recombinant Human DNASE in Cystic Fibrosis Patients With Chronic Sinusitis to Prevent Acute Sinusitis Exacerbations and Improve Symptoms and Outcomes - A Pilot Study
Brief Title: Pulmozyme in Cystic Fibrosis With Sinusitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Never funded
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Timothy Craig, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#33344
Record Dates: First submitted 2010-06-25; First posted 2010-07-02 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2012-11

CONDITIONS: Sinusitis; Cystic Fibrosis
Keywords: sinusitis; cystic fibrosis; therapy
MeSH Terms: conditions — Sinusitis; Cystic Fibrosis | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PULMOZYME (Experimental): active drug
  Interventions: Drug: Pulmozyme single use ampule
- placebo (Placebo Comparator): cross over to placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pulmozyme single use ampule — • Each Pulmozyme single use ampule delivers 2.5 mL (2.5 mg) of the sterile solution to the nebulizer bowl. The aqueous solution contains 1.0 mg/mL dornase alfa, 0.15 mg/mL calcium chloride dihydrate, and 8.77 mg/mL sodium chloride.
  Other Names: Dornase alfa recombinant human deoxyribonuclease I (rhDNase)
  Arms: PULMOZYME
Drug: placebo — identical placebo
  Arms: placebo

SUMMARY:
The hypothesis is that the intranasal use of Pulmozyme will decrease the severity of sinusitis in Cystic Fibrosis and lead to an improved quality of life.

DETAILED DESCRIPTION:
The study will be a prospective enrollment of patients with CF and rhinosinusitis in a double-blind crossover study with nasal nebulized DNASE versus saline. Nebulization will be accomplished with PARI SinuStar nasal aerosol system nebulizer set powered by an air compressor. This will be a pilot study with each subject serving as their own control. Each arm of the study will be 3 months and randomization to active drug versus placebo will be generated without the knowledge of subject or researchers. A health care provider not involved in the care of the subject will be responsible for medication distribution and the randomization scheme. A daily diary will collect data for analysis. Visits will be arranged every 4 weeks at which time drug will be dispensed, adherence to daily diary and compliance to medication will be assessed. At each visit the SF-12, SNOT-20, Epworth Sleepiness Scale, Rhinitis Severity Scale, Nocturnal Rhinoconjunctivitis Quality of Life Specific Questionnaire (NRQLQ), Cystic Fibrosis Questionnaire-Revised, and Rhinosinusitis Quality of Life Survey will be utilized for acquisition of data (17-23). In addition, a Physician Global Assessment and a self administered patient rhinosinusitis VAS score (0-100 with 100 full recovery and 0 no effect) will be completed at each visit. To obtain objective data patients will have nasal endoscopic assessment at 4 different time points and nasal polyps and sinusitis rated on a scale as defined by Lund and Kennedy in the Ann Otol Laryngol 1995;104 (suppl 167):17-21. (24) Serial sinus CT scans will be avoided to decrease irradiation risk.

Subjects: A total of 12 patients will be enrolled in this pilot study, and recruitment will be through the Cystic Fibrosis Center at Penn State University, after IRB approval. All subjects must be over the age of 15 years (the age the investigators consider to be necessary to understand the consent and questionnaires required for the study), be of either gender and of any ethnicity. Subjects will be able to continue all presently used nasal and respiratory medications as long as the present therapeutic regimen has been used for one month prior to enrollment and these therapies have been used at a stable dose, method of distribution and without adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Patients with CF, age >15yo
2. Chronic sinusitis with symptoms
3. VAS score of at least 60 (0 to 100) reflecting symptoms associated with rhinosinusitis
4. CT scan demonstrating non-complicated sinusitis (defined as rhinosinusitis without orbit perforation, osteomyelitis, peri-sinus cellulitis, or meningitis)

Exclusion Criteria:

1. No evidence of sinusitis
2. VAS score for rhinosinusitis less than 60 on a scale of 0 to 100
3. Complicated sinusitis (defined as orbit perforation, osteomyelitis, peri-sinus cellulitis, meningitis complicating sinusitis)
4. Prior adverse events or allergy to DNASE
5. Unwilling to sign an approved IRB consent
6. Immediate indication for sinus surgery
7. Inability to adhere to therapy and understand and to complete questionnaires.
8. Being pregnant will exclude a subject from participating and the subjects will be requested to take birth control methods if actively engaging in sex. Further more, subjects will be requested to inform the investigators if they become pregnant. Pregnancy test will be performed at screening.
9. Active nursing of an infant will be an exclusion.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
1. To assess changes in quality of life of patients with Cystic Fibrosis while on DNASE as compared to placebo. | weeks
  Sinusitis will be a significant burden for patients with CF. Use of nasal nebulized recombinant human DNASE will demonstrate positive changes in symptoms of rhinosinusitis and will improve the quality of life of patients with Cystic Fibrosis. In addition, subjects on active therapy will have a decrease in acute infections and a decrease in disease burden as compared to when the subject is on placebo therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Craig, DO, Principal Investigator — Penn State University
Locations (1):
- Penn State Unicersity, Hershey, Pennsylvania, United States